CLINICAL TRIAL: NCT06418347
Title: Effect of Alpha-Lipoic Acid Supplementation on Polycystic Ovary Syndrome Clinical Outcome in Infertile Females Treated With Letrozole
Brief Title: Effect of ALA Combined With Letrozole on Polycystic Ovary Syndrome Clinical Outcome in Infertile Females
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALA on PCOS
Record Dates: First submitted 2024-03-29; First posted 2024-05-17 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-03

CONDITIONS: Polycystic Ovary Syndrome; Infertility, Female
Keywords: PCOS; ALA; Letrozole; Infertility; Ovulation rate
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility, Female; Infertility | interventions — Thioctic Acid; Letrozole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Other): This group will include 75 PCOS participants who will receive the standard treatment letrozole and the other commonly provided PCOS care (lifestyle modification, diet and exercise education, any other non-pharmacological method of management) according to the PCOS guidelines .Treatment with letrozole will begin after the baseline visit and for three cycles.
  Interventions: Drug: Letrozole
- Intervention (Experimental): this will include 75 PCOS participants who will receive the standard treatment as letrozole with the same schedule of the control group and the other commonly provided PCOS care as previously described in addition to ALA, (Thiotacid®, EVAPHARMA, Egypt) in a dose of one tablet "600 mg" three times per day Each patient in the test group will start the ALA from day 3 of the menstrual period then daily until the day of human chorionic gonadotropin (HCG) injection
  Interventions: Drug: Alpha lipoic acid; Drug: Letrozole

INTERVENTIONS:
Drug: Alpha lipoic acid — Alpha-lipoic acid (ALA), also known as 1,2-dithiolane-3-pentanoic acid or thioctic acid, is found in the mitochondria. It acts as an enzymatic cofactor for various enzymes in the Kreb's cycle. ALA has many beneficial properties making it a potential candidate for various clinical disorders. It is considered the universal or "ideal" antioxidant as it is both water-soluble and fat-soluble facilitating its passage across membran. ALA has direct as well as indirect anti-inflammatory effects. Being a potent antioxidant leads to a reduction in oxidative stress which in turn reduces inflammation, meaning ALA indirectly has anti-inflammatory effects. To add to ALA's benefits, it has anti-inflammatory properties that are independent of its antioxidant effects.
  Other Names: ALA
  Arms: Intervention
Drug: Letrozole — Letrozole is an aromatase inhibitor that controls the conversion of androgen to estrogen and increases ovarian androgens. The administration of letrozole in the follicular phase removes the effect of negative estrogen feedback on the pituitary and hypothalamus, thus increasing the gonadotropins]. When Letrozole blocks estrogen production, it encourages the body to produce more follicle-stimulating hormone (FSH).The additional FSH stimulates egg development and increases the likelihood of ovulation. Kar, S. Found that letrozole has excellent pregnancy rates compared to clomiphene citrate, Letrozole should be considered at par with clomiphene citrate as first-line drug for ovulation induction in infertile PCOS women.

SUMMARY:
This research study aims to investigate the effect of adding Alpha lipoic acid (ALA) supplement to letrozole treatment in infertile women with polycystic ovary syndrome (PCOS). The study will include 150 PCOS participants seeking fertility treatment. They will be randomly divided into two groups - control and intervention. Both groups will receive standard PCOS care including lifestyle counseling. The control group will be treated with letrozole only. The dose will start at (2.5 mg) for 5 days and can increase up to (7.5 mg) based on response. The intervention group will take ALA supplements along with letrozole treatment. ALA tablets (600mg) will be given three times daily starting from day 3 of the menstrual cycle till human chorionic gonadotropin (HCG) injection day. Letrozole dose for the intervention group will also follow the same incremental protocol as the control group. Patient monitoring will involve trans-vaginal ultrasound scans on certain cycle days to check follicle growth and the thickness of uterus lining. Once a follicle reaches 18mm in size, an intramuscular HCG injection will be given. Couples will be asked to have intercourse 36 hours after the injection.

Pregnancy will be tested two weeks later if menstruation does not occur. Metabolic, hormonal, and ultrasound parameters will be recorded at baseline and follow-ups. All adverse effects of the treatment will be noted. The study period will be a maximum of 3 treatment cycles or untill pregnancy is achieved. Outcome measures include ovulation and pregnancy rates. The effect of ALA on metabolic parameters (fasting glucose, fasting insulin, BMI and HOMA-IR), hormone levels (mid-luteal progesterone and serum estradiol), and follicular growth will also be assessed. Proper sample size and randomization methods will be followed. A Statistical analysis of collected data will help determine if ALA has additional benefits when combined with letrozole for PCOS fertility treatment. Finally, the results will be statistically analyzed. Statistical analysis will be done using the SPSS statistical software package.

DETAILED DESCRIPTION:
Eligible participants will be randomly allocated to the control group or the intervention group with a ratio of 1:1 after obtaining informed consent.

The two study groups will be as follows:

Control group: this group will include 75 PCOS participants who will receive the standard treatment letrozole and the other commonly provided PCOS care (lifestyle modification, diet and exercise education, any other non-pharmacological method of management) according to the PCOS guidelines.

Treatment with letrozole will begin after the baseline visit, and for three cycles, the administration will start after a spontaneous or progesterone-induced menstruation. In the first cycle, "2.5" mg letrozole will be taken for 5 days starting from day 3 to 7 of the menses, if no pregnancy was detected, letrozole dose will be increased to "5 mg" in the next cycle, and finally, "7.5 mg" letrozole will be administered during the third cycle if the patient is still unable to conceive.

Interventional group: this will include 75 PCOS participants who will receive the standard treatment as letrozole with the same schedule as the control group and the other commonly provided PCOS care as previously described in addition to ALA, (Thiotacid®, EVAPHARMA, Egypt) in a dose of one tablet "600 mg" three times per day Each patient in the test group will start the ALA from day 3 of the menstrual period, then daily until the day of human chorionic gonadotropin (HCG) injection.

Baseline assessment:

After enrollment, baseline data and demographics will be obtained from each participant including:

* Age and body mass index will be calculated in Kg/m^2.
* Serum FSH, LH, TSH, prolactin, androgens, including free and total testosterone and SHBG.
* Ultrasound measurements including antral-follicles count and detection of Polycystic ovaries "defined as either 12 or more follicles measuring 2 to 9 mm in diameter or an increased ovarian volume >10 cm^3.".
* Menstrual cyclicity, presence of first degree relatives with diabetes mellitus , smoking status, comorbidities, medication history .
* All subjects will be educated about their diet and physical activity, and they will be asked not to start any new medications during the study without informing the principal investigator.

Patients monitoring and follow-up. All the participants included in the study after a spontaneous or progesterone-induced menstrual cycle will be randomly assigned to either Control group or Interventional group and will be monitored by trans-vaginal ultrasound to assess follicular diameter and endometrial thickness on the 10th day of the cycle, then on 12th , 14th and the 20th days of the cycle for assessment of dominant follicle ( ≥ 18 mm) on TVUS. The number of dominant follicles and the endometrial thickness will be documented for each menstrual cycle.

* When at least one dominant follicle is detected, participants will receive an intramuscular injection of 10 000 IU human chorionic gonadotropin (HCG) (Choriomon, IBSA).
* An HCG injection will be given when at least one follicle measuring at least 18 mm is observed.
* Ovulation will also be confirmed by the evaluation of serum progesterone each cycle between cycle days 20-22 ( > 5 ng/mL) and the test will be repeated 1 week later if the initial progesterone level is below the threshold to confirm ovulation.
* Couples will be instructed to have timed intercourse 36 hours after the HCG injection.
* Serum HCG will be determined 2 weeks after HCG injection in the absence of menstruation for the detection of pregnancy.
* Pregnant women will be required to stop all medication.
* Patients who do not have any dominant follicles, will start a new ovulation induction cycle in the following month.
* Treatment of the next cycle will start if menses occurs either spontaneously or by induction. The first day of the menses is considered the first day of the cycle and this is repeated for up to a total of 3 treatment cycles.
* For those who fail to achieve a dominant follicle, alpha lipoic acid will be stopped and restarted in the next cycle as before.

ELIGIBILITY:
Inclusion Criteria:

* Female patient aged 18-35
* Willing to conceive
* PCOS, diagnosed according to the revised 2003 Rotterdam consensus criteria. " Oligo- or anovulation secondary to PCOS and at least one of the remaining two criteria: hyperandrogenism or polycystic ovarian morphology on ultrasound .
* Anovulation and/or infertility ≥ 1 year.
* At least one patent fallopian tube
* Normal uterine cavity
* Male partner with sperm concentration of at least 14 million/mL in at least one ejaculate.

Exclusion Criteria:

* Other causes for the infertility (male factor, tubal factor).
* Intake of hormonal or other drugs that can potentially influence the ovulation.
* Causes of anovulation or hyperandrogenism other than PCOS such as uncontrolled thyroid dysfunction or hyperprolactinemia.
* Contraindication to pregnancy
* Myo-inositol use < 3 months prior to study enrollment
* Concomitant metformin use. Previous use is allowed with last use at least 6 weeks prior to randomization.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is cumulative ovulation rate | 1 year
  which is defined as the proportion of cycles in which ovulation occurred in the whole follow-up period.

SECONDARY OUTCOMES:
The clinical pregnancy rate | 1 year
  ultrasound visualization of one or more gestational sac with pulsating fetal pole
BMI in kg/m^2 | 1 year
  weight in kilograms, height in meters will be combined to report BMI in kg/m^2
HOMA-IR | 1 year
  fasting insulin in (microU/L), fasting glucose in (nmol/L) will be combined to report HOMA-IR
serum estradiol | 1 year
  Will be measure in (pg/ml)
mid-luteal progesterone | 1 year
  Will be measured in (pg/ml)
size of follicles | 1 year
  Will be measured in (mm)
number of dominant follicles (≥18 mm) | 1 year
  Number of mature follicles in each ovary.
endometrial thickness | 1 year
  Will be measured in (mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fruzzetti F, Benelli E, Fidecicchi T, Tonacchera M. Clinical and Metabolic Effects of Alpha-Lipoic Acid Associated with Two Different Doses of Myo-Inositol in Women with Polycystic Ovary Syndrome. Int J Endocrinol. 2020 Mar 19;2020:2901393. doi: 10.1155/2020/2901393. eCollection 2020. PMID 32256570
- [Background] Genazzani AD, Shefer K, Della Casa D, Prati A, Napolitano A, Manzo A, Despini G, Simoncini T. Modulatory effects of alpha-lipoic acid (ALA) administration on insulin sensitivity in obese PCOS patients. J Endocrinol Invest. 2018 May;41(5):583-590. doi: 10.1007/s40618-017-0782-z. Epub 2017 Oct 31. PMID 29090431
- [Background] Masharani U, Gjerde C, Evans JL, Youngren JF, Goldfine ID. Effects of controlled-release alpha lipoic acid in lean, nondiabetic patients with polycystic ovary syndrome. J Diabetes Sci Technol. 2010 Mar 1;4(2):359-64. doi: 10.1177/193229681000400218. PMID 20307398